

## **Parental Consent Form**

Chief Investigator: Julie Johnson

Principal Investigator:

[We recommend you use an electronic consent form if you do not require any personal identifying information – see electronic consent form]

GUEP/NICR Approval Number [8017]

Participant number [Insert]

**Research Project Title:** The Breakfast Rise, Education and Knowledge study in children and young people who have Type 1 Diabetes (T1D): The BREAK study.

| | Please initial | box |
|---|---|---|
| 1 | I confirm that I have read and understood the Participant Information Sheet for parents/carers dated 08/10/2022 | |
| | version 2 explaining the above research project and I have had the opportunity to ask questions about the project. | |
| 2 | I understand that my child's participation is voluntary and that my child is free to withdraw at any time during the | |
| | study without giving a reason, and without any penalty. I understand that data collected up to the point of | |
| | withdrawal will still be used in the study. | |
| 3 | I understand that my child's responses will be kept anonymous using the participant number and I give permission | |
| | for members of the research team to have access to my child's anonymised responses. | |
| 4 | I give permission for my child's Healthcare professional to collect information about my child from my child's | |
| | medical records and that this will be shared with the research team. | |
| 5 | I agree for research data collected in the study to be given to the researchers, I understand that any data that leave | |
| | the research group will be fully anonymised so that my child cannot be identified. | |
| 6 | I understand that my child's General Practitioner (GP) will NOT be informed of my participation in this study. I | |
| | understand my child's diabetes team will be informed. If the researcher has any concerns regarding information | |
| | about my child and any measurements that are taken as part of this research, I will be advised to contact my | |
| | diabetes team or GP. | |
| 7 | I give permission for the research team to see my child's CGM readings for the duration of this study | |
| 8 | I understand that my child's personal data (your email address, their date of birth and the artificial identifiers) will | |
| | be kept for 6-12 months after the end of the study. | |
| 9 | I agree for my child to take part in this study. | |

| Name | of I | Parti | cip | ant |
|------|------|-------|-----|-----|
|------|------|-------|-----|-----|

| Name of Parent consenting | Signature: |
|---------------------------|------------|

Date: Click here to enter a date

Date: Click here to enter a date

Name of Principal Investigator Signature:

Date: Click here to enter a date

When completed: 1 for parent, 1 for Principal Investigator site file, 1 to be filed in medical notes, 1 for Chief Investigator